CLINICAL TRIAL: NCT06868888
Title: The Effect of Osmotic Stress in Erythrocyte Rheology in ESRD Patients
Brief Title: Rheological Functions of Erythrocyte in ESRD
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jong-Shyan Wang, Professor, Chang Gung Memorial Hospital
Other Study IDs: 202102279A3102
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: End-stage Renal Disease (ESRD)
Keywords: Hemodialysis; Aerobic capacity; Deformability; Erythrocyte
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Blood Specimen Collection; Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ESRD: ESRD patients under hemodialysis
  Interventions: Other: Blood collection; Other: Cardiopulmonary exercise testing (CPET)
- Health control: Healthy sedentary volunteers
  Interventions: Other: Blood collection; Other: Cardiopulmonary exercise testing (CPET)

INTERVENTIONS:
Other: Blood collection — Erythrocyte osmotic deformability was evaluated via osmotic gradient ektacytometry.
Other: Cardiopulmonary exercise testing (CPET) — Cardiopulmonary Exercise Testing (CPET) is a non-invasive assessment that evaluates the integrated function of the cardiovascular, pulmonary, and muscular systems during exercise.

SUMMARY:
End-stage renal disease (ESRD) disrupts erythrocyte deformability due to osmotic imbalances, oxidative stress, and uremic toxins, leading to impaired microcirculation and oxygen transport. Dysregulation of ion channels, particularly the Gardos channel, exacerbates dehydration and eryptosis, further compromising vascular integrity. Given the critical role of erythrocyte flexibility in oxygen delivery, this study investigates its relationship with aerobic capacity in ESRD patients, highlighting potential mechanisms of microvascular dysfunction

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) profoundly alters osmotic homeostasis, disrupting erythrocyte deformability and impairing microcirculatory dynamics, ultimately compromising oxygen delivery to tissues. Persistent oxidative stress, hyperosmotic fluctuations, and accumulation of uremic toxins collectively modulate ion channel activity, particularly by stimulating cation influx and perturbing calcium regulation. These disruptions accelerate erythrocyte aging and promote eryptosis, a programmed form of red blood cell death. Furthermore, dysregulation of the Gardos channel exacerbates potassium efflux, leading to excessive cell dehydration, increased blood viscosity, and further deterioration of vascular integrity. Given the pivotal role of erythrocyte flexibility in oxygen transport efficiency, impairments in osmotic deformability may contribute to the reduced aerobic capacity frequently observed in ESRD patients. This study aims to elucidate the interplay between erythrocyte biomechanical properties and cardiopulmonary fitness in this population, shedding light on potential therapeutic targets to mitigate microvascular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Receiving hemodialysis and medication at least for 6 weeks
* Kt/V score > 1.2

Exclusion Criteria:

* Under 20 years-old
* Hyperkalemia occurs within 3 month
* Having orthopedic or muscular diseases
* Other concerned medical, psychological or physiological diseases
* Pregnancy
* Other exercise contraindications

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study included 18 patients with end-stage renal disease (ESRD) and 18 age-matched healthy controls. ESRD patients were recruited and with inclusion criteria requiring a confirmed diagnosis of ESRD and stable dialysis treatment for at least three months. Healthy controls were free of chronic illnesses and were matched by age and sex. Exclusion criteria included a history of hyperkalemia within the past three months, heart failure, pregnancy, or any condition contraindicating cardiopulmonary exercise testing. All participants underwent assessments within one week of enrollment, and written informed consent was obtained before participation."
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-03-26 (Estimated)

PRIMARY OUTCOMES:
Deformability of erythrocytes | Data collection was completed within one week of participant enrollment
  Deformability refers to the cells' ability to adapt their shape to the dynamically changing flow conditions so as to minimize their resistance to flow.
Aggregation of erythrocytes | Data collection was completed within one week of participant enrollment
  Erythrocyte aggregation is the reversible clumping of red blood cells (RBCs) under low shear forces or at stasis.
Cardiopulmonary fitness | Data collection was completed within one week of participant enrollment
  ESRD patients performed cardiopulmonary exercise testing (CPET) to assess their aerobic capacity. CPET composed of continuous workload increment of 10 W/min until exhaustion (usually within 8-12 minutes). Oxygen consumption, carbon dioxide production, ventilation, respiratory rate would be recorded.

SECONDARY OUTCOMES:
Quality of life in ESRD patients | Data collection was completed within one week of participant enrollment
  The investigators would use a qusionnaire, The Kidney Disease Quality of Life 36-item short form survey (KDQOL-36), to record and scale the qulaity of life in ESRD patients. The KDQOL-36 (Kidney Disease Quality of Life 36-Item Short Form Survey) measures the quality of life in kidney disease patients. It uses a score range from 0 to 100, where higher scores indicate better quality of life and lower scores indicate worse outcomes. Ensure to note this when reporting results to clarify that higher scores reflect fewer symptoms and better overall well-being.
Gardos function | Data collection was completed within one week of participant enrollment
  Gardos channel activation leads to K⁺ efflux, followed by water loss, resulting in erythrocyte dehydration and increased fragility. Dysfunctional regulation of this channel contributes to impaired microcirculation and reduced oxygen delivery, exacerbating vascular complications in ESRD.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No